CLINICAL TRIAL: NCT07002541
Title: NOL-Guided Intraoperative Remifentanil Consumption With PECS-II and Erector Spinae Plane Blocks in Breast Surgery: A Randomized Controlled Trial
Brief Title: PECS-II vs ESP in Nociception Level Index Guided Breast Surgery
Acronym: NOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Associate professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024.424.IRB1.047
Record Dates: First submitted 2025-05-07; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Intraoperative Pain; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PECS-II group (Active Comparator)
  Interventions: Procedure: PECS II block
- ESP group (Active Comparator)
  Interventions: Procedure: ESP block
- Control group (No Intervention)

INTERVENTIONS:
Procedure: PECS II block — The PECS-II block is an ultrasound-guided interfascial plane block designed to provide analgesia for surgeries involving the anterolateral chest wall, particularly breast surgery. It is an extension of the PECS-I block, which targets the medial and lateral pectoral nerves. In the PECS-II technique, a high-frequency linear ultrasound probe is used to identify the fascial planes. A 22G, 50 mm regional block needle is advanced in-plane under sterile conditions. A total of 30 mL of 0.25% bupivacaine is administered: 10 mL is injected between the pectoralis major and minor muscles (targeting the pectoral nerves), and 20 mL between the pectoralis minor and serratus anterior muscles (to block the lateral branches of intercostal nerves and intercostobrachial nerve).
  Arms: PECS-II group
Procedure: ESP block — The erector spinae plane (ESP) block is a fascial plane block performed under ultrasound guidance to provide multimodal analgesia for thoracic and abdominal surgeries, including breast procedures. In this technique, a high-frequency linear ultrasound probe is used to visualize the transverse process of the thoracic vertebra, typically at the T4-T5 level. With the patient in a seated position and under standard sterile conditions, a 22G, 50 mm regional block needle is inserted in-plane until the tip reaches the fascial plane between the erector spinae muscle and the transverse process. After negative aspiration, 1-2 mL of test dose is injected to confirm correct needle placement by observing separation of fascial layers. Then, 20 mL of 0.25% bupivacaine is injected incrementally.
  Arms: ESP group

SUMMARY:
Background:

Breast surgery is often associated with significant perioperative pain. While systemic opioids are commonly used, their side effects (nausea, vomiting, respiratory depression, delayed recovery) have encouraged the adoption of regional anesthesia techniques for better analgesia and reduced opioid requirements. PECS-II and Erector Spinae Plane (ESP) blocks are two effective regional techniques frequently utilized in breast surgery. However, comparative data on their impact on intraoperative opioid consumption under nociception-guided anesthesia remains limited.

The Nociception Level Index (NOL) is an objective monitoring tool that integrates multiple physiological signals (e.g., heart rate variability, skin conductance, pulse amplitude) to assess nociceptive responses in real-time. When used intraoperatively, it enables more precise opioid titration, potentially optimizing analgesia while minimizing opioid exposure.

Objective:

To compare the efficacy of PECS-II and ESP blocks in reducing intraoperative remifentanil consumption during breast surgery under general anesthesia guided by NOL monitoring.

Methods:

This prospective, randomized controlled trial was conducted at Koç University Hospital following ethical approval. Ninety female patients aged 18-80 years, classified as ASA I-III and scheduled for elective mastectomy or other breast surgeries, were randomly assigned into three groups (n=30 each):

Group 1 (PECS-II Block) Group 2 (ESP Block) Group 3 (Control - no block) Regional blocks were performed before surgery with ultrasound guidance. PECS-II block was administered at the 3rd to 5th rib levels in the mid-axillary line using 30 mL of 0.3% bupivacaine. ESP block was applied at T2-T5 levels with a total of 20 mL 0.5% bupivacaine.

All patients received standardized general anesthesia, including propofol, fentanyl, rocuronium, and desflurane maintenance. Remifentanil infusion (0.05-0.1 μg/kg/min) was titrated based on NOL values every 5 minutes: increased by 0.03 μg/kg/min if NOL >25, and decreased by 0.03 μg/kg/min if NOL <10.

Data collected included:

Total intraoperative remifentanil consumption (primary outcome) NOL scores every 5 minutes Postoperative pain scores (NRS) at 1st, 6th, 12th, and 24th hours (at rest and with arm abduction) Total opioid consumption (morphine, tramadol) in the first 24 hours Opioid-related side effects (nausea, vomiting, pruritus) Length of hospital stay Blinding was applied to data collectors (pain nurses and anesthesia technicians), but due to the nature of the procedures, surgeons and anesthesiologists were not blinded.

Statistical Analysis:

Data were analyzed using SPSS v26. Continuous variables were tested for normality (Shapiro-Wilk), and analyzed with t-tests or Mann-Whitney U as appropriate. Categorical variables were compared using Chi-square tests. Significance was set at p<0.05.

Expected Outcomes and Contribution:

It is hypothesized that both PECS-II and ESP blocks will significantly reduce intraoperative remifentanil consumption compared to the control group. Furthermore, these blocks may improve postoperative pain control, reduce opioid-related side effects, and shorten recovery time.

This study aims to clarify the relative efficacy of two widely used regional blocks in the context of objective, nociception-guided anesthesia. The findings are expected to support evidence-based use of regional techniques in breast surgery and contribute to the growing body of literature emphasizing opioid-sparing strategies in perioperative care.

ELIGIBILITY:
Eligibility Criteria This study involves adult female patients undergoing elective breast surgery for benign or malignant conditions. The goal is to evaluate the effectiveness of regional anesthesia techniques (PECS-II and ESP blocks) in reducing intraoperative opioid consumption, guided by Nociception Level Index (NOL) monitoring.

Inclusion Criteria:

Female patients aged 18 to 80 years ASA Physical Status Classification I-III

Scheduled for elective unilateral or bilateral breast surgery, including one or more of the following:

Lumpectomy with axillary lymph node biopsy or dissection Breast reconstruction Breast reduction Mastopexy Implant expander removal or placement

Exclusion Criteria:

Morbid obesity (BMI > 40 kg/m²) Presence of non-sinus cardiac rhythm Chronic opioid use (defined as daily use for >2 weeks in the last month or total use >4 weeks) History of opioid abuse or dependence Comorbidities causing moderate to severe functional limitation Inability to communicate with study personnel or follow instructions Pregnancy or breastfeeding Known allergy or hypersensitivity to bupivacaine or any study-related medication

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative remifentanyl consumption | The time frame for intraoperative remifentanil consumption refers to the entire duration of the surgical procedure, starting from skin incision to the end of surgery (skin closure).

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes